CLINICAL TRIAL: NCT01084291
Title: A Phase I Evaluation of the Safety and Immunogenicity of the rDEN1∆30 Dengue Serotype 1 Vaccine Given at a Single Dose of 101 PFU in Healthy Flavivirus-naïve Adult Subjects
Brief Title: Evaluation of the Safety and Immune Response to an Investigational Dengue Type 1 Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIR 253
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Dengue Virus
Keywords: Vaccine; Dengue Hemorrhagic Fever
MeSH Terms: conditions — Severe Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DEN1 Vaccine (Experimental): Participants will receive a single dose of investigational vaccine for dengue virus subtype 1.
  Interventions: Biological: Investigational Vaccine for DEN1
- Placebo (Placebo Comparator): Participants will receive a single dose of placebo vaccine.
  Interventions: Other: Placebo injection

INTERVENTIONS:
Biological: Investigational Vaccine for DEN1 — Subcutaneous injection in upper arm of vaccine at dose of 10 plaque-forming units (PFU)
  Other Names: rDEN1∆30 vaccine
  Arms: DEN1 Vaccine
Other: Placebo injection — Subcutaneous injection of placebo
  Arms: Placebo

SUMMARY:
Dengue viruses can cause dengue fever and other serious health conditions, primarily affecting people living in tropical regions of the world. There are four types of dengue virus, and infection with one does not offer protection against the others. This study will test whether a vaccine developed to prevent infection with dengue virus type 1 (DEN1) causes a response in people's immune system and is safe.

DETAILED DESCRIPTION:
The dengue virus causes approximately 50 million cases of dengue fever and 1.5 million cases of the more severe diseases dengue hemorrhagic fever (DHS) and dengue shock syndrome (DSS) every year. There are four subtypes of the virus, and infection with one offers no protection from infection by the others. In fact, most cases of DHS and DSS occur in people infected by more than one subtype. In areas of the world where multiple subtypes of dengue are common, vaccines must be developed against each of the subtypes of dengue virus. This study will examine the safety and immune response of an investigational vaccine for preventing infection with DEN1.

Participation in this study will last about 6 weeks. Participants will be randomly assigned to be injected with either the investigational study vaccine or a placebo. Participants will have a five in six chance of receiving the vaccine. The first study visit will take place on the vaccination day, on which participants will undergo a physical examination, blood draw, and pregnancy test, and then receive the vaccine. Participants will be given a thermometer and temperature card, and be told to record their temperature three times per day for 16 days after vaccination. Participants will come to follow-up visits every other day for the 16 days after vaccination, and then 3, 4, and 6 weeks after vaccination (Days 21, 28, and 42). Assessments completed during these visits will include a questionnaire about how the participant is feeling, pregnancy test, review of temperature cards, blood draw, and physical exam. Blood drawn will be analyzed to check participants' health, determine the amount of vaccine and antibodies in the blood, test markers in white blood cells and genes, and look for proteins that are important for fighting dengue infection.

ELIGIBILITY:
Inclusion Criteria:

* In good general health as determined by physical examination, laboratory screening, and review of medical history
* Available for the duration of the study, including approximately 6 weeks post-vaccination
* Female participants of childbearing potential must be willing to use effective contraception for the duration of the trial

Exclusion Criteria:

* Currently breast-feeding or pregnant
* Exhibits evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies
* Presence of a behavioral, cognitive, or psychiatric disease that affects the ability of the participant to understand and cooperate with the requirements of the study protocol
* Has screening laboratory values of Grade 1 or above for absolute neutrophil count (ANC), ALT, and serum creatinine, as defined in this protocol
* Presence of any condition that would jeopardize the safety or rights of the participant or would render the participant unable to comply with the protocol
* Significant alcohol or drug abuse in the past 12 months which has caused medical, occupational, or family problems, as indicated by participant history
* History of a severe allergic reaction or anaphylaxis
* Severe asthma (emergency room visit or hospitalization within the last 6 months)
* Presence of HIV infection, determined by screening and confirmatory assays
* Presence of hepatitis C virus (HCV) infection, determined by screening and confirmatory assays
* Presence of hepatitis B virus (HBV) infection, determined by hepatitis B surface antigen (HBsAg) screening
* Presence of any known immunodeficiency syndrome
* Uses anticoagulant medications
* Has used corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 42 days prior to or following vaccination. An immunosuppressive dose of corticosteroids is defined as greater than or equal to 10 mg prednisone equivalent per day for greater than or equal to 14 days.
* Has received a live vaccine within 28 days or a killed vaccine within 14 days prior to vaccination or anticipated receipt of any vaccine during the 42 days following vaccination
* Has no spleen
* Received blood products within the past 6 months, including transfusions or immunoglobulin or anticipated receipt of any blood products or immunoglobulin during the 42 days following vaccination
* History or serologic evidence of previous dengue virus infection or other flavivirus infection (e.g., yellow fever virus, St. Louis encephalitis, West Nile virus)
* Has received a flavivirus vaccine (licensed or experimental)
* Anticipates receipt of any investigational agent in the 42 days before or after vaccination
* Participant has definite plans to travel to a dengue endemic area during the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-04; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related adverse events (AEs), as classified by both severity and seriousness, through active and passive surveillance | Measured throughout study
Immunogenicity to dengue virus subtype one (DEN1), as assessed by neutralizing antibody titers | Measured 4 and 6 weeks after vaccination

SECONDARY OUTCOMES:
Frequency, quantity, and duration of viremia following vaccination | Measured every other day after vaccination for 16 days, and on Days 21, 28, and 42
Number of vaccinees infected with DEN1, defined as recovery of vaccine virus from the blood or serum of a participant and/or by seroconversion to DEN1 | Measured at study completion
Comparison of the infectivity rates, safety, and immunogenicity of a single dose of DEN1 vaccine to those rates of previous clinical trials | Measured at study completion

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — CIR, Johns Hopkins University; Beth Kirkpatrick, MD, Principal Investigator — University of Vermont
Locations (2):
- United States (2):
  - Fletcher Allen Health Care (FAHC) General Clinical Research Center (GCRC), Burlington, Vermont
  - University of Vermont Vaccine Testing Center, Burlington, Vermont

REFERENCES:
- [Background] Blaney JE Jr, Durbin AP, Murphy BR, Whitehead SS. Development of a live attenuated dengue virus vaccine using reverse genetics. Viral Immunol. 2006 Spring;19(1):10-32. doi: 10.1089/vim.2006.19.10. PMID 16553547
- [Background] Whitehead SS, Falgout B, Hanley KA, Blaney JE Jr, Markoff L, Murphy BR. A live, attenuated dengue virus type 1 vaccine candidate with a 30-nucleotide deletion in the 3' untranslated region is highly attenuated and immunogenic in monkeys. J Virol. 2003 Jan;77(2):1653-7. doi: 10.1128/jvi.77.2.1653-1657.2003. PMID 12502885